CLINICAL TRIAL: NCT03411096
Title: Comparison of Analgesic Efficacy of Quadratus Lumborum Block With Local Anesthesia and Quadratus Lumborum Block With Placebo Only After Ileostomy Repair: a Randomized, Double-blind, Non-inferiority Trial
Brief Title: Quadratus Lumborum Block : Local Anesthesia Versus Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Soo Yeun Park, Principal Investigator, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KNUHC02
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Loop Ileostomy; Colorectal Disorders
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus lumborum block (Experimental): Quadratus lumborum block with 0.75% ropivacaine
  Interventions: Procedure: Quadratus lumborum block using ropivacaine
- Placebo (Placebo Comparator): Quadratus lumborum block with normal saline
  Interventions: Procedure: Quadratus lumborum block with normal saline

INTERVENTIONS:
Procedure: Quadratus lumborum block using ropivacaine — After general anesthesia, an anesthesiologist will perform an quadratus lumborum block with 0.75% ropivacaine (20cc) under ultrasound guidance.
  Other Names: Quadratus lumborum block
  Arms: Quadratus lumborum block
Procedure: Quadratus lumborum block with normal saline — After general anesthesia, an anesthesiologist will perform an quadratus lumborum block with normal saline (20cc) under ultrasound guidance.
  Arms: Placebo

SUMMARY:
Opioid analgesics have many side effects. Quadratus lumborum (QL) block is one kind of regional nerve block that can reduce the side effects of opioid analgesics. The investigators hypothesize that QL block with local analgesics (ropivacaine) can significantly reduce pain intensity in comparison with placebo.

DETAILED DESCRIPTION:
Opioid analgesics have been used to control the pain. However, many postoperative complication, such as nausea, vomiting, constipation, ileus, etc are related to opioid usage. Recently, local or regional pain nerve block, such as transversus abdominis plane block, wound infiltration, have been reported in several studies. Quadratus lumborum (QL) block was first introduced in the abstract of 2007 European Society of Regional Anesthesia. The effect is longer and more than that of transversus abdominis plane block because it works close to the spinal cord nerves. The QL block can be an effective pain control method for patients who underwent ileostomy closure. The aim of this study is to compare pain intensity after ileostomy closure between QL block (ropivacaine) group and placebo group (normal saline).

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-75 years, either sex
* Patients scheduled to undergo elective ileostomy repair surgery under general anesthesia.
* Patients underwent curative surgery and ileostomy due to colorectal cancer.
* Willingness and ability to sign an informed consent document

Exclusion Criteria:

* Allergies to anesthetic or analgesic medications
* Contraindication to the use of locoregional anesthesia
* Chronic opioid use
* Coagulopathy, Impaired kidney function, uncontrolled diabetes, psychiatric disorders, severe cardiovascular impairment or chronic obstructive lung disease
* Necessity of major resection other than colorectal, palliative surgery
* BMI above 35kg/m2
* American Society of Anesthesiologists (ASA) physical status above 3

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pain numerical rating scale (NRS) | 6 hours after surgery
  1. Pain NRS during rest and cough
  2. NRS scale 0-10:0, "no pain"; 10, "worst pain imaginable"

SECONDARY OUTCOMES:
Pain NRS | 2, 12,24,36,48,72 hour after surgery
  1. Pain NRS during rest and cough
  2. NRS scale 0-10:0, "no pain"; 10, "worst pain imaginable"
Rescue opioid analgesic requirement | postoperative day 0,1,2,3
  Overall postoperative rescue of opioid analgesic requirement described by using the Defined Daily Dose
Postoperative nausea and vomiting scale | 2, 12,24,36,48,72 hour after surgery
  Postoperative nausea and vomiting scores (assessed using a 0-2 categorical scale; no nausea/nausea/vomiting)
Occurrence of prolonged post-operative ileus | 8 weeks after surgery
  Occurrence of prolonged post-operative ileus (assessed using a 0-1 categorical scale; no ileus/ ileus)
Time to first oral fluid intake | 8 weeks after surgery
  Time to first oral fluid intake after surgery
Time to first oral soft diet | 8 weeks after surgery
  Time to first oral soft diet after surgery
Length of hospital stay | 8 weeks after surgery
  Length of hospital stay after admission

CONTACTS AND LOCATIONS:
Overall Officials: Jin Seok Yeo, MD, Study Director — Kyungpook National University Chilgok Hospital; In Teak Woo, MD, Study Chair — Kyungpook National University Chilgok Hospital; Soo Yeun Park, MD, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Chilgok Hospital, Daegu, South Korea